CLINICAL TRIAL: NCT01198600
Title: Ocular Comfort and the "Aging" Lens (ERBIUM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-373-C-006
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-07

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1: Habitual no Replacement, then Habitual Replacement (Other): Contact lenses per participant's habitual prescription worn for 30 days with no replacement, followed by contact lenses per habitual prescription worn for 30 days with a replacement pair dispensed at Day 28.
  Interventions: Device: Habitual contact lens
- Phase 1: Habitual Replacement, then Habitual no Replacement (Other): Contact lenses per participant's habitual prescription worn for 30 days with replacement pair dispensed at Day 28, followed by contact lenses per habitual prescription worn for 30 days with no replacement.
  Interventions: Device: Habitual contact lens
- Phase 2: Lotrafilcon B Replacement (Other): Contact lenses worn for 56 days with replacement pair dispensed at Day 28.
  Interventions: Device: Lotrafilcon B contact lens; Device: Contact lens cleaning and disinfecting system (ClearCare)
- Phase 3: Lotrafilcon B Replacement Replacement (Other): Contact lenses worn for 43 days with replacement pair dispensed at Day 1 and Day 28.
  Interventions: Device: Lotrafilcon B contact lens; Device: Contact lens cleaning and disinfecting system (ClearCare)

INTERVENTIONS:
Device: Habitual contact lens — Hydrogel or silicone hydrogel contact lens per participant's habitual brand and prescription
  Arms: Phase 1: Habitual Replacement, then Habitual no Replacement; Phase 1: Habitual no Replacement, then Habitual Replacement
Device: Lotrafilcon B contact lens — Commercially marketed silicone hydrogel contact lens
  Other Names: AIR OPTIX AQUA
  Arms: Phase 2: Lotrafilcon B Replacement; Phase 3: Lotrafilcon B Replacement Replacement
Device: Contact lens cleaning and disinfecting system (ClearCare) — Commercially marketed, hydrogen peroxide-based contact lens care system
  Other Names: CLEARCARE
  Arms: Phase 2: Lotrafilcon B Replacement; Phase 3: Lotrafilcon B Replacement Replacement

SUMMARY:
The purpose of this trial was to evaluate the factors affecting comfortable contact lens wear and how those factors affect contact lens replacement frequency.

DETAILED DESCRIPTION:
Eligible participants began Phase 1, following either Cycle A or Cycle B, and crossing over to the second cycle after completing the first. After the Phase 1 results were evaluated, eligible participants entered Phase 2. After Phase 2 results were evaluated, participants who consistently reported the highest and the lowest comfort scores entered Phase 3 and were defined as either survivors or strugglers.

ELIGIBILITY:
Inclusion Criteria:

* At least 17 years of age.
* Ocular exam in the last two years.
* Currently wearing hydrogel or silicone hydrogel contact lenses on a daily wear basis with a monthly replacement schedule.
* Wearing contact lenses at least five days per week for a minimum of 10 hours each day.
* Able to wear lenses in the available power range with a best-corrected visual acuity of at least 20/32 in both eyes.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular disease.
* Systemic condition that may affect a study outcome.
* Using any systemic or topical medications that may affect ocular health.
* Wears lenses on an extended or continuous wear schedule.
* Habitually wears multifocal lenses.
* Other protocol-defined exclusion criteria may apply.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, MOptom FAAO, Study Director — University of Waterloo Centre for Contact Lens Research
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one Canadian research center.
Pre-assignment Details: Baseline characteristics are presented for all enrolled participants: 78. The participant flow chart includes all enrolled and dispensed participants: 72. Six participants were enrolled but not dispensed.
Groups:
- Phase 1: Habitual no Replacement, Then Habitual Replacement: Contact lenses per participant's habitual prescription worn for 30 days with no replacement, followed by contact lenses per habitual prescription worn for 30 days with a new pair dispensed at Day 28.
- Phase 1: Habitual Replacement, Then Habitual no Replacement: Contact lenses per participant's habitual prescription worn for 30 days with a new pair dispensed at Day 28, followed by contact lenses per habitual prescription worn for 30 days with no replacement.
- Phase 3: Lotrafilcon B Replacement Replacement: Contact lenses worn for 43 days with replacement pair dispensed on Day 1 and Day 28.
Period: Phase 1: Period One, 30 Days of Wear
Arm/Group | Phase 1: Habitual no Replacement, Then Habitual Replacement | Phase 1: Habitual Replacement, Then Habitual no Replacement | Phase 2: Lotrafilcon B Replacement | Phase 3: Lotrafilcon B Replacement Replacement
Started | 35 | 37 | 0 | 0
Completed | 33 | 36 | 0 | 0
Not Completed | 2 | 1 | 0 | 0
Not completed — Inconvenience | 1 | 0 | 0 | 0
Not completed — Asymptomatic infiltrates | 1 | 0 | 0 | 0
Not completed — Unable to achieve acceptable comfort | 0 | 1 | 0 | 0
Period: Phase 1: Period Two, 30 Days of Wear
Arm/Group | Phase 1: Habitual no Replacement, Then Habitual Replacement | Phase 1: Habitual Replacement, Then Habitual no Replacement | Phase 2: Lotrafilcon B Replacement | Phase 3: Lotrafilcon B Replacement Replacement
Started | 32 (One participant discontinued between Period One and Period Two due to unconvenience.) | 36 | 0 | 0
Completed | 32 | 35 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Inconvenience | 0 | 1 | 0 | 0
Period: Phase 2: 56 Days of Wear
Arm/Group | Phase 1: Habitual no Replacement, Then Habitual Replacement | Phase 1: Habitual Replacement, Then Habitual no Replacement | Phase 2: Lotrafilcon B Replacement | Phase 3: Lotrafilcon B Replacement Replacement
Started | 0 | 0 | 67 | 0
Completed | 0 | 0 | 62 | 0
Not Completed | 0 | 0 | 5 | 0
Not completed — Inconvenience | 0 | 0 | 2 | 0
Not completed — Relocation | 0 | 0 | 2 | 0
Not completed — Unable to achieve satisfactory comfort | 0 | 0 | 1 | 0
Period: Phase 3: 43 Days of Wear
Arm/Group | Phase 1: Habitual no Replacement, Then Habitual Replacement | Phase 1: Habitual Replacement, Then Habitual no Replacement | Phase 2: Lotrafilcon B Replacement | Phase 3: Lotrafilcon B Replacement Replacement
Started | 0 | 0 | 0 | 38
Completed | 0 | 0 | 0 | 38
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed participants.
Arm/Group | Overall
Number analyzed (Participants) | 78
Age Continuous [Mean (Standard Deviation); unit: years] | 25.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 13
Region of Enrollment [Number; unit: participants]
  Canada | 78

OUTCOME MEASURES:

1. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 1 Day, Hour 1
Description: Ocular comfort was rated bilaterally by the participant after wearing the same pair of lenses for 1 day. Ocular comfort was recorded on a continuum and converted to a 100-point scale where 1=EXTREMELY UNCOMFORTABLE ("I CANNOT tolerate the comfort of my eyes! I am in pain!")and 100=VERY COMFORTABLE & FRESH ("Wow! My eyes feel incredible! I love this feeling.")
Time Frame: Day 1
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Survivors: Lotrafilcon B/Replacement/Replacement: Contact lenses worn for 43 days, with initial dispense on Day 0 and subsequent dispenses on Days 1 and 15 during Phase 3. "Survivors" were participants who reported no or very little reduction in subjective comfort between Day 1 and Day 27 of Phase 2.
- Strugglers: Lotrafilcon B/Replacement/Replacement: Contact lenses worn for 43 days during Phase 3, with initial dispense on Day 0 and subsequent dispenses on Days 1 and 15. "Strugglers" were participants who reported a reduction in subjective comfort of at least 15 points on a 100-point scale between Day 1 and Day 27 of Phase 2.
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 76 (14) | 88 (14)

2. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 1 Day, Hour 10
Description: as for outcome 1
Time Frame: Day 1
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Survivors: Lotrafilcon B/Replacement/Replacement: Contact lenses worn for 43 days during Phase 3, with initial dispense on Day 0 and subsequent dispenses on Days 1 and 15. "Survivors" were participants who reported no or very little reduction in subjective comfort between Day 1 and Day 27 of Phase 2.
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 69 (19) | 76 (19)

3. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 1 Day, End of Day
Description: as for outcome 1
Time Frame: Day 1
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 65 (21) | 67 (21)

4. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 14 Days, Hour 1
Description: Ocular comfort was rated bilaterally by the participant after wearing the same pair of lenses for 14 days. Ocular comfort was recorded on a continuum and converted to a 100-point scale where 1=EXTREMELY UNCOMFORTABLE ("I CANNOT tolerate the comfort of my eyes! I am in pain!")and 100=VERY COMFORTABLE & FRESH ("Wow! My eyes feel incredible! I love this feeling.")
Time Frame: Day 15
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Strugglers: Lotrafilcon B/Replacement/Replacement: Contact lenses worn for 43 days during Phase 3, with initial dispense on Day 0 and subsequent dispenses on Days 1 and 15. "Strugglers" were participants who reported a reduction in subjective comfort of at least 15 points on a 100-point scale between Day 1 and Day 27 of Phase 2.of Phase 2.
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 80 (14) | 79 (14)

5. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 14 Days, Hour 10
Description: as for outcome 4
Time Frame: Day 15
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 77 (19) | 64 (19)

6. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 14 Days, End of Day
Description: as for outcome 4
Time Frame: Day 15
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 72 (21) | 60 (21)

7. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 27 Days, Hour 1
Description: Ocular comfort was rated bilaterally by the participant after wearing the same pair of lenses for 27 days. Ocular comfort was recorded on a continuum and converted to a 100-point scale where 1=EXTREMELY UNCOMFORTABLE ("I CANNOT tolerate the comfort of my eyes! I am in pain!")and 100=VERY COMFORTABLE & FRESH ("Wow! My eyes feel incredible! I love this feeling.")
Time Frame: Day 43
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 78 (14) | 74 (14)

8. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 27 Days, Hour 10
Description: as for outcome 7
Time Frame: Day 43
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 72 (19) | 63 (19)

9. Primary Outcome: Phase 3: Ocular Comfort, Lens Age 27 Days, End of Day
Description: as for outcome 7
Time Frame: Day 43
Population: All enrolled and dispensed participants, Phase 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Survivors: Lotrafilcon B/Replacement/Replacement | Strugglers: Lotrafilcon B/Replacement/Replacement
Number analyzed (Participants) | 22 | 16
Units on a scale | 66 (21) | 57 (21)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 8-JUL-2010 to 19-JUL-2011.
Description: The safety population includes all enrolled and dispensed participants.
Groups:
- Habitual Contact Lens: Contact lens per participant's habitual prescription worn for two 30-day periods in Phase 1, with a replacement dispensed at Day 28 in either Period 1 or Period 2.
- Lotrafilcon B Contact Lens: Contact lens worn for 56 days with a replacement dispensed at Day 28 in Phase 2, followed by 43 days in Phase 3 with a replacement dispensed at Day 1 and Day 14.
Arm/Group | Habitual Contact Lens | Lotrafilcon B Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/67
Other Adverse Events (participants affected / at risk) | 0/78 | 0/67

LIMITATIONS AND CAVEATS:
The current study design and sample size was not able to uncover clinically meaningful differences between survivors and strugglers. There is considerable individual variation in lens performance with age, which requires further investigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.